CLINICAL TRIAL: NCT06869499
Title: Niemann-PID: Study of the Prevalence of Acid Sphingomyelinase Deficiency/Niemann Pick AB and B Disease in Patients With Diffuse Interstitial Lung Disease
Brief Title: Study of the Prevalence of Acid Sphingomyelinase Deficiency/Niemann Pick AB and B Disease in Patients With Diffuse Interstitial Lung Disease
Acronym: Niemann-PID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wladimir MAUHIN, Dr (Other)
Collaborators: Bichat Hospital (Other); Hospital Avicenne (Other); Rennes University Hospital (Other); Bicetre Hospital (Other); University Hospital, Marseille (Other); Tenon Hospital, Paris (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Lille (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor-Investigator, Wladimir MAUHIN, Dr, Internist, Groupe Hospitalier Diaconesses Croix Saint-Simon
Organization: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-A00050-47
Record Dates: First submitted 2025-02-19; First posted 2025-03-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: Splenomegaly; Splenectomy; Thrombopenia; Interstitial Lung Disease (ILD); Hypocholesterolemia
Keywords: Acid sphingomyelinase deficiency; Ground glass lesions; Niemann Pick A/B, B; lysoSM; smpd1; splenomegaly; interstitial lung disease; screening; acid sphingomyelinase
MeSH Terms: conditions — Splenomegaly; Thrombocytopenia; Lung Diseases, Interstitial; Niemann-Pick Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This study is a multicenter prospective interventional research involving humans with minimal risks and constraints.
  The minimal risks and study add-ons are:
  -4ml blood sample for acid sphingomyelinase enzyme activity and LysoSM, if required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Cohort (Experimental): The participants will be asked for a :
  1. Venous blood collection (4ml EDTA tube) for the determination of :
     * acid sphingomyelinase enzyme activity in all participants included in the study. The determination of acid sphigomyelinase enzyme activity will be performed using a multiplex blotting assay that allows simultaneous determination of acid sphigomyelinase activity (ASMD) by tandem MS/MS mass spectrometry, but also Beta-glucocerebrosidase (Gaucher disease), alpha-galactosidase (Fabry disease), Maltase Acid (Pompe disease), Galactocerebrosidase (Krabbe disease), Alpha-L iduronidase (control enzyme) (MPSI)).
     * if acid sphingomyelinase activity < 1.82 μmol/h/l (decreased) is detected, the concentration of lysoSM should be determined on the same sample.
  2. Appropriate participant care management in the event of a positive ASMD screening.
  Interventions: Procedure: Blood sampling for dosage

INTERVENTIONS:
Procedure: Blood sampling for dosage — 4ml blood sample to measure acid sphingomyelinase enzyme activity and LysoSM, if required.

SUMMARY:
The goal of this clinical trial is to optimise and facilitate screening for Acid SphingoMyelinase Deficiency (ASMD) disease, by evaluating acid sphingomyelinase activity and, where appropriate, LysoSM levels in a cohort of 200 participants with diffuse interstitial lund disease (ILD) at risk of developing ASMD disease.

ILD is common in the general population, so in order to limit the number of differential diagnoses, the population to be studied will be restricted to participants aged between 15 years and 3 months and 60 years, with ILD plus ground-glass opacities on chest CT scan certified by a pulmonologist/radiologist or internist, AND splenomegaly or splenectomy, and/or thrombocytopenia, and/or low HDL cholesterol, and/or parental consanguinity which increase the sensitivity of ASMD screening.

In this clinical trail, two procedures are added, participants will be asked for :

* a blood sample to measure the acid sphingomyelinase enzyme activity and LysoSM, if required.
* a follow-up visit at 6 months

DETAILED DESCRIPTION:
With the prevalence of ASMD estimated to be between 0.4 and 0.6/100,000 births, is probably under-diagnosed because it is not well known. Based on the current literature, no prevalence studies have been carried out, particularly in patients with interstitial lung disease (ILD). Similarly, no decision-making algorithm has been established for screening for ASMD in this participant population. Therefore, we aim to conduct this multicenter clinical trial to assess the relevance of implementing a decision algorithm to optimise screening for ASMD. Validation of this algorithm could provide clinicians with an additional diagnostic tool to improve the management of this disease and prevent its progression. Olipudase-alfa, a specific treatment for ASMD available from 2022, could thus benefit a greater number of people with disease who have been under-diagnosed.

The literature reports an association between chronic visceral ASMD (type B) and the presence of ILD, usually accompanied by splenomegaly or splenectomy (whatever the medical reason or cause), low HDL cholesterol, thrombocytopenia, with a higher frequency in cases of parental consanguinity.

ILD is common in the general population, therefore, in order to limit the number of differential diagnoses, the population to be studied will consist of participants aged between 15 years and 3 months and 60 years, with diffuse interstitial lung disease with ground-glass opacities on chest CT scan certified by a pulmonologist/radiologist or internist. We will propose acid sphingomyelinase activity testing in this population in case of splenomegaly (palpable spleen or craniocaudal length ≥ 13 cm) or splenectomy and/or thrombocytopenia (platelets < 150 G/L) and/or low HDL cholesterol (<0.4 g/l or 1. 03 mmol/l) and/or parental consanguinity increase the sensitivity of ASMD screening.

Considering that detection of ASMD after the age of 60 would not lead to a modification in current management, it was decided to limit the population to 60 years of age. Screening for ASMD, a very rare disease, can only be reasonably performed in a limited and selected population.

Description of actions and procedures added by the research :

* Venous blood collection (4ml EDTA tube) for the determination of :

  * acid sphingomyelinase enzyme activity in all participants included in the study. The determination of acid sphigomyelinase enzyme activity will be performed using a multiplex blotting assay that allows simultaneous determination of acid sphigomyelinase activity (ASMD) by tandem MS/MS mass spectrometry, but also Beta-glucocerebrosidase (Gaucher disease), alpha-galactosidase (Fabry disease), Maltase Acid (Pompe disease), Galactocerebrosidase (Krabbe disease), Alpha-L iduronidase (control enzyme) (MPSI)).
  * if acid sphingomyelinase activity < 1.82 μmol/h/l (decreased) is detected, the concentration of lysoSM should be determined on the same sample.
* Appropriate participant management in the event of a positive ASMD screening.

ELIGIBILITY:
Inclusion Criteria:

1. Interstitial lung disease with ground-glass lesions on a chest CT scan certified by a pneumologist/radiologist or internist.
2. At least one of the following criteria :

   * Splenomegaly (palpable spleen or craniocaudal length ≥ 13 cm)
   * Splenectomy
   * Thrombocytopenia (platelets < 150 G/L)
   * Low HDL-cholesterol (<0.4 g/l or 1.03 mmol/l)
   * Notion of parental consanguinity
3. Have given their written informed consent, in accordance with regulations.
4. Affiliated to the social security system or entitled beneficiary (excluding AME).

Exclusion Criteria:

1. Inability to understand the information provided.
2. Under guardianship, curatorship or legal protection.
3. Under restraint or deprived of liberty by judicial or administrative decision.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Optimising screening for ASMD in a population of adult patients with diffuse interstitial pneumopathy | 12 months
  To optimise and facilitate screening for ASMD by evaluating acid sphingomyelinase activity and, where appropriate, LysoSM levels in a cohort of 200 patients with diffuse interstitial pneumopathy disease at risk of developing ASMD.

CONTACTS AND LOCATIONS:
Overall Officials: Wladimir MAUHIN, Doctor, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided